CLINICAL TRIAL: NCT01400386
Title: Bioavailability of Chlorogenic and Phenolic Acids From Soluble Coffees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 10.04.Met
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Soluble coffee 1 (Experimental)
  Interventions: Other: Coffee bioavailability trial
- Soluble coffee 2 (Experimental)
  Interventions: Other: Coffee bioavailability trial
- Soluble coffee 3 (Experimental)
  Interventions: Other: Coffee bioavailability trial
- Soluble coffee 4 (Experimental)
  Interventions: Other: Coffee bioavailability trial

INTERVENTIONS:
Other: Coffee bioavailability trial — Coffee bioavailability trial

SUMMARY:
Coffee contributes to a large extent to our daily intake of phenolic compounds which have been associated with potential health benefits. A study by Richelle et al. (2001), using an LDL oxidation assay, showed that phenolic compounds in coffee possessed antioxidant activity which varied depending on the coffee bean source and the degree of roasting. Little is known about the bioavailability of phenolic compounds from coffee at various roasting degrees. Therefore, further human studies are required in order to demonstrate the absorption, and bioavailability of metabolites that may also be efficient in vivo.

The main objective of this clinical trial is to investigate the possible difference in the bioavailability of chlorogenic and phenolic acids from coffee at various roasting levels.

DETAILED DESCRIPTION:
Coffee contributes to a large extent to our daily intake of phenolic compounds which have been associated with potential health benefits. A study by Richelle et al. (2001), using an LDL oxidation assay, showed that phenolic compounds in coffee possessed antioxidant activity which varied depending on the coffee bean source and the degree of roasting. Little is known about the bioavailability of phenolic compounds from coffee at various roast levels. Therefore, further human studies are required in order to demonstrate the absorption, and bioavailability of metabolites that may also be efficient in vivo.

The main objective of this clinical trial is to investigate the possible difference in the bioavailability of chlorogenic and phenolic acids from coffee at different roast levels.

After medical examination and approval, subjects will be randomly assigned to one of the four coffee treatments. Each study period correspond to the ingestion of one the treatments and study periods are separated by a one week washout period. Blood will be taken as a time course for 24h while urine will be collected for 30h. Investigators are also blinded with respect to the dose and the treatment given to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 60 years, male and female
* healthy as determined by the medical questionnaire and the medical visit
* normal weight: BMI 19 - 25
* Coffee drinkers with an average consumption of 2-5 cups per day
* having given informed consent

Exclusion Criteria:

* Intestinal or metabolic diseases / disorders such as diabetic, renal, hepatic, hypertension, pancreatic or ulcer
* food allergy
* Have had a major gastrointestinal surgery
* Difficulty to swallow
* Have a regular consumption of medication
* Have taken antibiotic therapy within the last 6 months
* Alcohol consumption > 2 units a day
* Smokers > 5 cigarettes a day
* Have given blood within the last 3 weeks before the start of the study
* Volunteers who cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial during the last 3 weeks

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetics: sum of AUC of chlorogenic and phenolic acids the of extreme treatments. | 18 months

SECONDARY OUTCOMES:
Composite of pharmacokinetics: AUC, Sum of AUC, Cmax, Tmax and T1/2 of plasma chlorogenic and phenolic acids from the other treatments. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, Ph.D, Principal Investigator — Société des Produits Nestlé (SPN)
Locations (1):
- NESTEC/Clinical Development Unit / Metabolic Unit, Lausanne, Canton of Vaud, Switzerland